CLINICAL TRIAL: NCT01015625
Title: Primary Operation in SYnchronous meTastasized InVasivE Breast Cancer, a Multicenter Prospective Randomized Study to Evaluate the Use of Local Therapy
Brief Title: Primary Operation in SYnchronous meTastasized InVasivE Breast Cancer
Acronym: POSYTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Bayer (Industry); Amgen (Industry); Hoffmann-La Roche (Industry); AstraZeneca (Industry); Sanofi (Industry); Wyeth-Lederle Pharma GmbH (Industry); GlaxoSmithKline (Industry); Merck Sharp & Dohme LLC (Industry); Fond of the Viennese Mayor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ABCSG 28 / POSYTIVE; ABCSG 28 (Other: ABCSG)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Synchronous Metastasized Breast Cancer; Circulating Tumor Cells
Keywords: breast cancer; ABCSG; POSYTIVE; growth factor; median survival; surgery on demand; surgical therapy; blood specimen; tissue specimen; VEGF; TGF; circulating tumor cells; stem cells
MeSH Terms: conditions — Neoplastic Cells, Circulating; Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Surgical Therapy (Other): Local therapy consists of lumpectomy or mastectomy with or without radiotherapy (according to center tumor board decision) with a resection free margin of at least 1 mm or more demonstrated on paraffin embedded histological sections. Intraoperative frozen sections are allowed but not definitive for margin assessment. Sentinel node biopsy may be performed and has always to be followed by axillary dissection of level I and II (axillary surgery level I and II is mandatory).
  Interventions: Procedure: Surgery
- B: Surgery on Demand (Other): In Arm B (no local therapy) it may be necessary to perform local therapy on demand (surgery, radiotherapy). Reasons may be uncontrolled bleeding or infected exulcerations with a septic component and no treatment benefit from conservative therapy. This will be considered as protocol deviation. However, the patient's follow up is recorded and data are available for analyses as intention to treat.
  Interventions: Procedure: Surgery on Demand

INTERVENTIONS:
Procedure: Surgery — lumpectomy or mastectomy with or without radiotherapy. Sentinel biopsy followed by axillary dissection (level I-II)
  Arms: A: Surgical Therapy
Procedure: Surgery on Demand — if necessary local therapy on demand
  Arms: B: Surgery on Demand

SUMMARY:
Primary Operation in synchronous metastasized invasive breast cancer to evaluate the use of local therapy

DETAILED DESCRIPTION:
This study is a prospective, randomized, multicentre, study concerning the influence of local treatment on the patients with synchronous metastasized breast cancer. Patients will be stratified at inclusion according to the centre, the menopausal status (pre-menopausal, post-menopausal), the hormone-receptor status (ER-/PR-/not determinable; any PR and/or Er+), the HER-2 status (positive vs. negative/not determinable), the grading (G1/G2/not determinable vs. G3), location of metastases (visceral ± vs bone only), organs with metastases (single organ vs multiple organs) and use of first line chemotherapy (anthracycline ± vs. taxane vs others). Thereafter patients will be randomly assigned to receive either local therapy of the breast (lumpectomy or mastectomy + axillary surgery /± radiotherapy) versus no local therapy. Systemic therapy will be administered at the centers policy.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years
* Eastern Cooperative Oncology Group Performance Status is 0 -2
* Untreated synchronous metastasized invasive carcinoma of the breast with the primary tumor in situ (bilateral synchronous metastasized breast cancer patients are eligible)
* The primary tumor must be identified and may be any size, however, primary resection with resection free margins must be possible
* Invasive adenocarcinoma of the breast on histological examination
* The metastatic site must be identified by radiological assessment(Computer Tomography of the chest and the abdomen OR ultrasound and chest x ray for visceral metastases; bone scan AND/OR computer tomography AND/OR magnetic resonance for bone metastases). A biopsy is not necessary.
* Written informed consent must be obtained and documented prior to beginning any protocol specific procedures and according to local regulatory requirements
* able to comply with the protocol requirements during the treatment and follow-up period.

Exclusion Criteria:

* Patients in whom a R0 resection (microscopic free margins) is clinically questionable
* Inflammatory cancer
* Patients with a brain metastasis
* Patients who are not eligible for general anesthesia and operations
* Patients without metastatic breast cancer (patients with a tumor marker value (CEA, CA15-3) above normal levels without the radiological proven evidence of metastases are not eligible for the study)
* Patients with a second untreated malignancy
* Any previous malignancy treated with curative intent and the patient has not been disease-free for 5 years - exceptions are: (a)carcinoma in situ of the cervix, (b)squamous carcinoma of the skin, (c)basal cell carcinoma of the skin
* Patients with any recurrent cancer disease
* Pregnant or lactating women
* Patients are not allowed to be part of another local therapy trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-11-24 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Fitzal, MD, Study Director — Austrian Breast & Colorectal Cancer Study Group; Michael Gnant, MD, Study Director — Austrian Breast & Colorectal Cancer Study Group; Guenther Steger, MD, Study Director — Austrian Breast & Colorectal Cancer Study Group
Locations (14):
- Austria (14):
  - Hospital Guessing, Güssing, Burgenland
  - Hospital Oberpullendorf, Oberpullendorf, Burgenland
  - Ordination Dr. Wette, Saint Veit A. D. Glan, Carinthia
  - Gynaegological Medical University Graz, Graz, Styria
  - Medical University Graz, Oncology, Graz, Styria
  - Medical University of Innsbruck, Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH - BHS Linz, Coop. Study Group, Linz, Upper Austria
  - Ordensklinikum Linz GmbH - Elisabethinen Linz, Linz, Upper Austria
  - General Hospital Linz, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
  - State Hospital Feldkirch, Feldkirch, Vorarlberg
  - Paracelsus Medical University Salzburg-Oncology, Coop. Group, Salzburg
  - Medical University of Vienna-General Hospital Vienna, Vienna
  - Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babiera GV, Rao R, Feng L, Meric-Bernstam F, Kuerer HM, Singletary SE, Hunt KK, Ross MI, Gwyn KM, Feig BW, Ames FC, Hortobagyi GN. Effect of primary tumor extirpation in breast cancer patients who present with stage IV disease and an intact primary tumor. Ann Surg Oncol. 2006 Jun;13(6):776-82. doi: 10.1245/ASO.2006.03.033. Epub 2006 Apr 17. PMID 16614878
- [Background] Blanchard DK, Bhatia P, Hilsenbeck SG, Elledge RM. Does surgical management of stage IV breast cancer effect outcome? SABCC 2006, San Antonio
- [Background] Carmichael AR, Anderson ED, Chetty U, Dixon JM. Does local surgery have a role in the management of stage IV breast cancer? Eur J Surg Oncol. 2003 Feb;29(1):17-9. doi: 10.1053/ejso.2002.1339. PMID 12559070
- [Background] Khan SA, Stewart AK, Morrow M. Does aggressive local therapy improve survival in metastatic breast cancer? Surgery. 2002 Oct;132(4):620-6; discussion 626-7. doi: 10.1067/msy.2002.127544. PMID 12407345
- [Background] Rapiti E, Verkooijen HM, Vlastos G, Fioretta G, Neyroud-Caspar I, Sappino AP, Chappuis PO, Bouchardy C. Complete excision of primary breast tumor improves survival of patients with metastatic breast cancer at diagnosis. J Clin Oncol. 2006 Jun 20;24(18):2743-9. doi: 10.1200/JCO.2005.04.2226. Epub 2006 May 15. PMID 16702580
- [Background] Gnerlich J, Jeffe DB, Deshpande AD, Beers C, Zander C, Margenthaler JA. Surgical removal of the primary tumor increases overall survival in patients with metastatic breast cancer: analysis of the 1988-2003 SEER data. Ann Surg Oncol. 2007 Aug;14(8):2187-94. doi: 10.1245/s10434-007-9438-0. Epub 2007 May 24. PMID 17522944
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Flanigan RC, Salmon SE, Blumenstein BA, Bearman SI, Roy V, McGrath PC, Caton JR Jr, Munshi N, Crawford ED. Nephrectomy followed by interferon alfa-2b compared with interferon alfa-2b alone for metastatic renal-cell cancer. N Engl J Med. 2001 Dec 6;345(23):1655-9. doi: 10.1056/NEJMoa003013. PMID 11759643
- [Background] Mickisch GH, Garin A, van Poppel H, de Prijck L, Sylvester R; European Organisation for Research and Treatment of Cancer (EORTC) Genitourinary Group. Radical nephrectomy plus interferon-alfa-based immunotherapy compared with interferon alfa alone in metastatic renal-cell carcinoma: a randomised trial. Lancet. 2001 Sep 22;358(9286):966-70. doi: 10.1016/s0140-6736(01)06103-7. PMID 11583750
- [Background] Norton L, Massague J. Is cancer a disease of self-seeding? Nat Med. 2006 Aug;12(8):875-8. doi: 10.1038/nm0806-875. No abstract available. PMID 16892025
- [Background] Al-Hajj M, Clarke MF. Self-renewal and solid tumor stem cells. Oncogene. 2004 Sep 20;23(43):7274-82. doi: 10.1038/sj.onc.1207947. PMID 15378087
- [Background] Bao S, Wu Q, McLendon RE, Hao Y, Shi Q, Hjelmeland AB, Dewhirst MW, Bigner DD, Rich JN. Glioma stem cells promote radioresistance by preferential activation of the DNA damage response. Nature. 2006 Dec 7;444(7120):756-60. doi: 10.1038/nature05236. Epub 2006 Oct 18. PMID 17051156
- [Background] Al-Hajj M, Wicha MS, Benito-Hernandez A, Morrison SJ, Clarke MF. Prospective identification of tumorigenic breast cancer cells. Proc Natl Acad Sci U S A. 2003 Apr 1;100(7):3983-8. doi: 10.1073/pnas.0530291100. Epub 2003 Mar 10. PMID 12629218
- [Background] Kong FM, Anscher MS, Murase T, Abbott BD, Iglehart JD, Jirtle RL. Elevated plasma transforming growth factor-beta 1 levels in breast cancer patients decrease after surgical removal of the tumor. Ann Surg. 1995 Aug;222(2):155-62. doi: 10.1097/00000658-199508000-00007. PMID 7543740
- [Background] Tang B, Vu M, Booker T, Santner SJ, Miller FR, Anver MR, Wakefield LM. TGF-beta switches from tumor suppressor to prometastatic factor in a model of breast cancer progression. J Clin Invest. 2003 Oct;112(7):1116-24. doi: 10.1172/JCI18899. PMID 14523048
- [Background] Yang YA, Dukhanina O, Tang B, Mamura M, Letterio JJ, MacGregor J, Patel SC, Khozin S, Liu ZY, Green J, Anver MR, Merlino G, Wakefield LM. Lifetime exposure to a soluble TGF-beta antagonist protects mice against metastasis without adverse side effects. J Clin Invest. 2002 Jun;109(12):1607-15. doi: 10.1172/JCI15333. PMID 12070308
- [Background] Kim KJ, Li B, Winer J, Armanini M, Gillett N, Phillips HS, Ferrara N. Inhibition of vascular endothelial growth factor-induced angiogenesis suppresses tumour growth in vivo. Nature. 1993 Apr 29;362(6423):841-4. doi: 10.1038/362841a0. PMID 7683111
- [Background] Linderholm B, Grankvist K, Wilking N, Johansson M, Tavelin B, Henriksson R. Correlation of vascular endothelial growth factor content with recurrences, survival, and first relapse site in primary node-positive breast carcinoma after adjuvant treatment. J Clin Oncol. 2000 Apr;18(7):1423-31. doi: 10.1200/JCO.2000.18.7.1423. PMID 10735889
- [Background] Linderholm BK, Lindh B, Beckman L, Erlanson M, Edin K, Travelin B, Bergh J, Grankvist K, Henriksson R. Prognostic correlation of basic fibroblast growth factor and vascular endothelial growth factor in 1307 primary breast cancers. Clin Breast Cancer. 2003 Dec;4(5):340-7. doi: 10.3816/cbc.2003.n.039. PMID 14715109
- [Background] Nishimura R, Nagao K, Miyayama H, Matsuda M, Baba K, Yamashita H, Fukuda M. Higher plasma vascular endothelial growth factor levels correlate with menopause, overexpression of p53, and recurrence of breast cancer. Breast Cancer. 2003;10(2):120-8. doi: 10.1007/BF02967636. PMID 12736564
- [Background] Wu Y, Saldana L, Chillar R, Vadgama JV. Plasma vascular endothelial growth factor is useful in assessing progression of breast cancer post surgery and during adjuvant treatment. Int J Oncol. 2002 Mar;20(3):509-16. PMID 11836562
- [Background] Kummel S, Eggemann H, Luftner D, Thomas A, Jeschke S, Zerfel N, Heilmann V, Emons G, Zeiser T, Ulm K, Kobl M, Korlach S, Schmid P, Sehouli J, Elling D, Blohmer JU. Changes in the circulating plasma levels of VEGF and VEGF-D after adjuvant chemotherapy in patients with breast cancer and 1 to 3 positive lymph nodes. Anticancer Res. 2006 Mar-Apr;26(2C):1719-26. PMID 16617567
- [Background] Caine GJ, Stonelake PS, Lip GY, Blann AD. Changes in plasma vascular endothelial growth factor, angiopoietins, and their receptors following surgery for breast cancer. Cancer Lett. 2007 Apr 8;248(1):131-6. doi: 10.1016/j.canlet.2006.06.011. Epub 2006 Aug 7. PMID 16891056
- [Background] Curigliano G, Petit JY, Bertolini F, Colleoni M, Peruzzotti G, de Braud F, Gandini S, Giraldo A, Martella S, Orlando L, Munzone E, Pietri E, Luini A, Goldhirsch A. Systemic effects of surgery: quantitative analysis of circulating basic fibroblast growth factor (bFGF), Vascular endothelial growth factor (VEGF) and transforming growth factor beta (TGF-beta) in patients with breast cancer who underwent limited or extended surgery. Breast Cancer Res Treat. 2005 Sep;93(1):35-40. doi: 10.1007/s10549-005-3381-1. PMID 16184456
- [Background] Joffe JK, Banks RE, Forbes MA, Hallam S, Jenkins A, Patel PM, Hall GD, Velikova G, Adams J, Crossley A, Johnson PW, Whicher JT, Selby PJ. A phase II study of interferon-alpha, interleukin-2 and 5-fluorouracil in advanced renal carcinoma: clinical data and laboratory evidence of protease activation. Br J Urol. 1996 May;77(5):638-49. doi: 10.1046/j.1464-410x.1996.09573.x. PMID 8689103
- [Background] Wagner JR, Walther MM, Linehan WM, White DE, Rosenberg SA, Yang JC. Interleukin-2 based immunotherapy for metastatic renal cell carcinoma with the kidney in place. J Urol. 1999 Jul;162(1):43-5. doi: 10.1097/00005392-199907000-00011. PMID 10379736
- [Background] Fitzal F, Sporn EP, Draxler W, Mittlbock M, Taucher S, Rudas M, Riedl O, Helbich TH, Jakesz R, Gnant M. Preoperative core needle biopsy does not increase local recurrence rate in breast cancer patients. Breast Cancer Res Treat. 2006 May;97(1):9-15. doi: 10.1007/s10549-005-6935-3. PMID 16502019
- [Background] El-Tamer MB, Ward BM, Schifftner T, Neumayer L, Khuri S, Henderson W. Morbidity and mortality following breast cancer surgery in women: national benchmarks for standards of care. Ann Surg. 2007 May;245(5):665-71. doi: 10.1097/01.sla.0000245833.48399.9a. PMID 17457156
- [Derived] Bjelic-Radisic V, Fitzal F, Knauer M, Steger G, Egle D, Greil R, Schrenk P, Balic M, Singer C, Exner R, Soelkner L, Gnant M; ABCSG. Primary surgery versus no surgery in synchronous metastatic breast cancer: patient-reported quality-of-life outcomes of the prospective randomized multicenter ABCSG-28 Posytive Trial. BMC Cancer. 2020 May 6;20(1):392. doi: 10.1186/s12885-020-06894-2. PMID 32375735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was randomized November 24, 2010, the last patient was randomized October 30, 2015. Randomization took place in 14 Austrian clinical sites. In total, 90 patients were enrolled.
Period: Overall Study
Arm/Group | A: Surgical Therapy | B: Surgery on Demand
Started | 45 | 45
Completed | 8 | 19
Not Completed | 37 | 26
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Death | 30 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Surgical Therapy | B: Surgery on Demand | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Full Range); unit: years] | 62 [23 to 85] | 65 [35 to 85] | 64 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
T-stage [Count of Participants; unit: Participants] — The clincial T-stage (cT) describes the categories of tumor size: cT1: <2 cm, cT2: 2 to 5 cm, cT3: > 5 cm, cT4: tumor has invaded other organs, like chest wall or skin.
  Participants
    cT1 | 11 | 7 | 18
    cT2 | 14 | 26 | 40
    cT3 | 10 | 3 | 13
    cT4 | 8 | 8 | 16
    Unkown | 2 | 1 | 3
N-stage [Count of Participants; unit: Participants] — The clinical N-stage describes the categories of affected lymph nodes: cN0: no lymph node affected, cN1: 1-3 lymph nodes affected, cN2: 4 to 9 lymph nodes affected, cN3: 10 or more lymph nodes affected.
  Participants
    cN0 | 10 | 10 | 20
    cN1 | 20 | 21 | 41
    cN2 | 7 | 2 | 9
    cN3 | 4 | 2 | 6
    Unknown | 4 | 10 | 14
Histologic grade [Count of Participants; unit: Participants] — The histologic grade describes to which extent the cancer cells and their arrangement look look like normal cells. Grade 1 (G1): well-differentiated, cells look more like normal breast tissue; Grade (G2): moderately differentiated; Grade (G3): poorly differentiated; GX: grade cannot be assessed.
  Participants
    G1 | 5 | 2 | 7
    G2 | 23 | 25 | 48
    G3 | 13 | 15 | 28
    Gx | 3 | 1 | 4
    Unknown | 1 | 2 | 3
Hormone receptor group [Count of Participants; unit: Participants]
  Estrogen and Progesterone negative | 9 | 8 | 17
  Any positive | 36 | 37 | 73
HER2 group [Count of Participants; unit: Participants]
  FISH amplified/IHC+++ | 10 | 8 | 18
  Negative | 35 | 36 | 71
  Unknown | 0 | 1 | 1
Surgery type [Count of Participants; unit: Participants]
  Breast-conserving | 12 | 3 | 15
  Modified radical | 30 | 4 | 34
  Missing | 3 | 38 | 41

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival with vs without local therapy (surgery)
Time Frame: Time from randomization until the last visit of the last participant; maximum time on study was 63.9 months
Population: Intent-to-treat population: All participants assigned to one of the two treatment arms were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Surgical Therapy | B: Surgery on Demand
Number analyzed (Participants) | 45 | 45
months | 34.6 [25.4 to 47.9] | 56.2 [34.0 to NA] — Not applicable, confidence limit cannot be calculated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: A: Surgical Therapy vs B: Surgery on Demand; To determine the effect of local therapy (surgery, Arm A) compared to systemic therapy only (Arm B) in synchronous metastasized breast cancer patients in terms of overall survival. Overall survival is defined as the time from randomization to death from any cause. Participants last known to be alive were censored at their last contact date or at the data cut-off date whichever came first; Test type: Superiority — A two-sided significance level of 5% was used; p = 0.042, Log Rank; Cox Proportional Hazard = 1.77, 95% CI 2-sided [1.01 to 3.09] — From the Cox Proportional hazard model with surgery vs no surgery fitted as a covariate. A hazard ratio > 1.0 indicates a higher average event rate and a shorter overall survival time for surgery relative to no surgery

2. Secondary Outcome: Time to Distant Progression
Description: Time to distant progression with vs without local therapy (surgery)
Time Frame: Time from randomization until the last visit of the last participant; maximum time on study was 63.9 months
Population: Intent-to-treat population: All participants assigned to one of the two treatment arms were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Surgical Therapy | B: Surgery on Demand
Number analyzed (Participants) | 45 | 45
months | 13.7 [5.9 to 20.0] | 24.4 [12.2 to 41.0]
Statistical Analysis 1: Comparison: A: Surgical Therapy vs B: Surgery on Demand; To determine the effect of local therapy (surgery) compared to systemic therapy only in synchronous metastasized breast cancer patients in terms of time from randomization to distant progression. Distant progression is defined as detection of new lesions or progression of existing metastases in locations different then breast. Participants last known to be alive without a distant progression were censored at their last contact date or at the data cut-off date whichever came first; Test type: Superiority — A two-sided significance level of 5% was used; p = 0.147, Log Rank; Cox Proportional Hazard = 1.45, 95% CI 2-sided [0.87 to 2.42] — From the Cox Proportional hazard model with surgery vs no surgery fitted as a covariate. A hazard ratio > 1.0 indicates a higher average event rate and a shorter time to distant progression for surgery relative to no surgery

3. Secondary Outcome: Time to Local Progression (TTPl)
Description: Time to local progression with vs without local therapy (surgery)
Time Frame: Time from randomization until the last visit of the last participant; maximum time on study was 63.9 months
Population: Intent-to-treat population: All participants assigned to one of the two treatment arms were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Surgical Therapy | B: Surgery on Demand
Number analyzed (Participants) | 45 | 45
months | 59.4 [43.1 to NA] — Not applicable, confidence limit cannot be calculated due to insufficient number of participants with events. | 55.8 [54.1 to NA] — Not applicable, confidence limit cannot be calculated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: A: Surgical Therapy vs B: Surgery on Demand; To determine the effect of local therapy (surgery) compared to systemic therapy only in synchronous metastasized breast cancer patients in terms of time from randomization to local progression. Local progression is defined as recurrence in breast with localization mamma, chest wall or axilla. Participants last known to be alive, who did not experience a local progression were censored at their last contact date or at the data cut-off date whichever came first; Test type: Superiority — A two-sided significance level of 5% was used; p = 0.890, Log Rank; Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.45 to 2.02] — From the Cox Proportional hazard model with surgery vs no surgery fitted as a covariate. A hazard ratio > 1.0 indicates a higher average event rate and a shorter time to local progression for surgery relative to no surgery

ADVERSE EVENTS:
Time Frame: Maximum observation period per patient for all-cause mortality was 10 years starting with randomization.
Description: All-cause mortality data presented for intention-to-treat analysis set and for the entire study. Serious adverse events and other (non-serious) adverse events were not assessed for the study.
Arm/Group | A: Surgical Therapy | B: Surgery on Demand
All-Cause Mortality (participants affected / at risk) | 30/45 | 22/45
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-02-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT01015625/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT01015625/SAP_001.pdf